CLINICAL TRIAL: NCT06506955
Title: An Open-label, Rollover Study of Futibatinib in Patients Previously Enrolled in an Antecedent Futibatinib Study
Brief Title: Futibatinib in Patients Previously Enrolled in an Antecedent Futibatinib as Monotherapy or Combination Therapy.
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS120-404
Record Dates: First submitted 2024-06-28; First posted 2024-07-18 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Advanced/Metastatic Cancer
Keywords: Futibatinib; TAS-120; FGFR; Cholangiocarcinoma; Breast cance; Urothelial Carcinom
MeSH Terms: conditions — Neoplasm Metastasis; Cholangiocarcinoma | interventions — futibatinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAS-120 (futibatinib) monotherapy (Experimental): TAS-120 tablets, oral, cycle length is defined as per antecedent study design
  Interventions: Drug: futibatinib
- TAS-120 (futibatinib) combination therapy with fulvestrant (Experimental): TAS-120 tablets in combination with fulvestrant, oral, cycle length is defined as per antecedent study design
  Interventions: Drug: futibatinib, fulvestrant

INTERVENTIONS:
Drug: futibatinib — TAS-120 futibatinib monotherapy
  Other Names: TAS-120
  Arms: TAS-120 (futibatinib) monotherapy
Drug: futibatinib, fulvestrant — TAS-120 futibatinib combination therapy with fulvestrant
  Other Names: TAS-120 + fulvestrant
  Arms: TAS-120 (futibatinib) combination therapy with fulvestrant

SUMMARY:
This is a nonrandomized, open-label, multicenter rollover study for patients who received futibatinib as monotherapy or as combination therapy in a Taiho-sponsored futibatinib study.

DETAILED DESCRIPTION:
TAS-120-404 is a nonrandomized, open-label, multicenter rollover study for patients who received futibatinib as monotherapy or as combination therapy in a Taiho-sponsored futibatinib study.

Patients who are still receiving futibatinib as monotherapy or as combination therapy, are deriving clinical benefit with no undue risk as assessed by the investigator, and have not met any of the antecedent protocol-specific discontinuation criteria are eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Receiving futibatinib as monotherapy or as combination therapy in an antecedent futibatinib study and deriving clinical benefit with no undue risk as assessed by the investigator.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test (urine or serum) within 7 days prior to receiving treatment. Both males and females of reproductive potential must agree to use effective birth control during study treatment and for a specified time after the last dose of study treatment.
* Ability to take medications orally (PO) (feeding tube is not permitted).

Exclusion Criteria:

• Has met any discontinuation criteria within the antecedent futibatinib study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with serious adverse events, treatment-related adverse events, and any AEs leading to treatment discontinuation graded according to NCI-CTCAE v5.0. | through study completion, an average of 5 years
  To collect long term safety information in patients continuing to receive treatment with futibatinib as monotherapy or in combination with fulvestrant who participated in a Taiho-sponsored futibatinib study and who are deriving clinical benefit with no undue risk

CONTACTS AND LOCATIONS:
Locations (9):
- University of California, San Francisco (UCSF), San Francisco, California, United States
- France (2):
  - Institut Paoli-Calmettes, Marseille
  - Institut De Cancerologie Strasbourg, Strasbourg
- Severance Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Universitari, Vall d'Hebron, Barcelona
  - Centro Integral Oncologico, Madrid
- United Kingdom (3):
  - Royal Marsden NHS Foundation Trust, London
  - Sarah Cannon Research Institute UK, London
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No